CLINICAL TRIAL: NCT06702202
Title: Comparison of the Effect of Subarachnoid Block and Femoropopliteal Block to Limb Perfusion in Patients with Peripheral Arterial Disease
Brief Title: Effect of Subarachnoid Block and Femoropopliteal Block to Limb Perfusion in PAD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes141124
Record Dates: First submitted 2024-11-14; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Arterial Disease; Subarachnoid Block; Femoropopliteal Block; Tissue Oxygen Saturation
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Femoropopliteal block (Group F) (Experimental): Ultrasonography was performed using the Mindray DP-10 system with a linear transducer positioned at the inguinal fold to identify and visualize the femoral nerve, 10 ml mixture of local anesthetics ( Marcaine® [bupivacaine HCl] 0,5% and Xylocaine® [Lidocaine HCL] 2% = 2:1) were injected in-plane around the femoral nerve. For popliteal sciatic nerve blocks, linear transducer was placed transversally on the distal thigh to visualize Sciatic nerve just before branching, followed by the injection of 20 ml of the same mixture of local anesthetics through a 50 mm block needle in-plane
  Interventions: Drug: Mixture of local anesthetics
- Subarachnoid block (Group S) (Experimental): Patients may assume either a sitting or lateral decubitus position, and subsequent to aseptic procedures, a G27 spinal needle will be introduced into the L3-4 interspinous space until clear cerebrospinal fluid visualization, followed by the injection of 2-2.5 ml of 0.5% hyperbaric Bupivacaine
  Interventions: Drug: 0.5% hyperbaric bupivacaine

INTERVENTIONS:
Drug: Mixture of local anesthetics — Marcaine® (bupivacaine HCl) 0,5% and Xylocaine® (Lidocaine HCL) 2% = 2:1 Given in Femoropopliteal block group (Group F)
  Arms: Femoropopliteal block (Group F)
Drug: 0.5% hyperbaric bupivacaine — Given in Subarachnoid block group (Group S)
  Arms: Subarachnoid block (Group S)

SUMMARY:
This pilot study investigates the effects of femoropopliteal and subarachnoid nerve blocks on tissue oxygen saturation (StO2) in patients with Peripheral Arterial Disease (PAD) during lower limb surgeries. Using Near-Infrared Spectroscopy (NIRS), the study compares changes in StO2 post-block. Although no significant differences were found between the two block types at most time points, subarachnoid blocks generally led to higher StO2 increases compared to femoropopliteal blocks, with significant differences observed at 5 and 15 minutes post-block.

DETAILED DESCRIPTION:
This pilot study explored the impact of femoropopliteal and subarachnoid nerve blocks on tissue oxygen saturation (StO2) in patients with Peripheral Arterial Disease (PAD) during lower limb surgeries, using Near-Infrared Spectroscopy (NIRS) for non-invasive monitoring. The study compared StO2 changes at baseline, 5, 15, and 30 minutes post-block in two groups: those receiving femoropopliteal blocks and those receiving subarachnoid blocks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old who are scheduled to undergo lower limb debridement surgery.
* Diagnosis of Peripheral Arterial Disease (PAD).
* Lesion located below the knee.

Exclusion Criteria:

* Consuming opioids before hospital admission.
* Having allergies to the medications used in the study.
* Presence of infection at the injection site.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Tissue Oxygen Saturation (StO2) | TI (Baseline): 10 minutes before the intervention; T2: 5 minutes after the intervention; T3: 15 minutes after the intervention; T4: 30 minutes after the intervention
  The primary outcome of this study is the percentage increase in tissue oxygen saturation (StO2) following the administration of femoropopliteal nerve blocks and spinal anesthesia. StO2 will be measured at two locations below the knee (Points A and B) at different heights. Measurements will be taken at four time points: 10 minutes before the intervention (TI), and 5, 15, and 30 minutes after the intervention (T2, T3, T4). The goal is to assess and compare the changes in StO2 induced by each type of anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No